CLINICAL TRIAL: NCT00345254
Title: Study That Clarifies Whether Cord Around the Neck Should be Severed at Delivery.
Brief Title: Severing Nuchal Cord at the Time of Delivery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Samuel Lurie, Professor, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS-SL-001
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Perinatal Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- severing cord (Experimental): The cord was cut intentionally after delivery of the anterior shoulder and prior to extraction of the body.
  Interventions: Procedure: severing cord
- Untouched cord (No Intervention): The cord was untouched after delivery of the anterior shoulder and prior to extraction of the body.

INTERVENTIONS:
Procedure: severing cord — The cord was cut intentionally after delivery of the anterior shoulder and prior to extraction of the body.
  Other Names: Cutting the umbilical cord
  Arms: severing cord

SUMMARY:
Umbilical cord often becomes encircled around portions of the fetus, usually the neck. The incidence ranges from 1 loop in 21% to 3 loops in 0.2%. In this study we wish to assessed the practice of severing the cord, which was encircled once around the neck of the fetus, after delivery of the anterior shoulder and prior to extraction of the body. The study and the control groups will include 30 women, each one. After diagnosis of cord around the neck during labor by ultrasound, the women will inter a randomization process. After delivery of the head, it will be cut intentionally in the study group and left intact in the control group. Neonatal outcome will be assessed.

DETAILED DESCRIPTION:
Umbilical cord often becomes encircled around portions of the fetus, usually the neck. The incidence ranges from 1 loop in 21% to 3 loops in 0.2%. In this study we wish to assessed the practice of severing the cord, which was encircled once around the neck of the fetus, after delivery of the anterior shoulder and prior to extraction of the body. The study and the control groups will include 30 women, each one. After diagnosis of cord around the neck during labor by ultrasound, the women will inter a randomization process. After delivery of the head, it will be cut intentionally in the study group and left intact in the control group. Neonatal outcome will be assessed.

ELIGIBILITY:
Inclusion Criteria:

single loop cord around the neck active labor spontaneous vaginal delivery

Exclusion Criteria:

instrumental delivery cesarean section false positive finding of cord around the neck multiple loop cord around the neck

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Sadan, MD, Principal Investigator — E Wolfson Medical Center, Holon, Israel
Locations (1):
- Deliveery Ward, Edith Wolfson Medical Center,, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severing Cord | Untouched Cord
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severing Cord | Untouched Cord | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Umbilical Cord pH
Time Frame: immediately after delivery
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Severing Cord | Untouched Cord
Number analyzed (Participants) | 30 | 30
pH | 7.29 (0.07) | 7.32 (0.06)
Statistical Analysis 1: Comparison: Severing Cord vs Untouched Cord; Test type: Superiority; p = 0.1, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Severing Cord | Untouched Cord
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes